CLINICAL TRIAL: NCT03050489
Title: AMIRI-CABG: Assessment of Myocardial Ischemic-Reperfusion Injury During Off- and On- Pump CABG
Brief Title: Assessment of Myocardial Ischemic-Reperfusion Injury During Off- and On- Pump CABG
Status: Completed | Type: Observational
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: AMIRI-CABG 03/17-11
Record Dates: First submitted 2017-02-06; First posted 2017-02-13 (Actual); Results first posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-04

CONDITIONS: Ischemic Heart Disease; Coronary Artery Disease; Ischemic Reperfusion Injury; CABG
Keywords: CABG; Off-Pump CABG; On-Pump CABG; ischemic-reperfusion injury during CABG; comparison of On- and Off- Pump CABG; Ischemic Heart Disease; Myocardial ischemia-reperfusion and myeloperoxidase; Myocardial ischemia-reperfusion biomarkers
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum from central vein.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- On-Pump CABG: Patients with coronary artery bypass graft (CABG) surgery performed with cardiopulmonary bypass.
  Interventions: Procedure: On-Pump CABG.
- Off-Pump CABG: Patients with coronary artery bypass graft (CABG) surgery performed without cardiopulmonary bypass.
  Interventions: Procedure: Off-Pump CABG.
- BH-CABG MSC.: Patients with coronary artery bypass graft (CABG) surgery performed on beating heart with mechanical support of circulation.
  Interventions: Procedure: BH-CABG MSC.

INTERVENTIONS:
Procedure: On-Pump CABG. — Standard On-Pump CABG.
  Groups: On-Pump CABG
Procedure: Off-Pump CABG. — Standard Off-Pump CABG.
  Groups: Off-Pump CABG
Procedure: BH-CABG MSC. — Patients with coronary artery bypass graft (CABG) surgery performed on beating heart with mechanical support of circulation
  Groups: BH-CABG MSC.

SUMMARY:
Assessment of myocardial ischemic-reperfusion injury during off- and on- pump CABG.

DETAILED DESCRIPTION:
Assessment of myocardial ischemic-reperfusion injury during off- and on- pump CABG is monitored by intraoperative measurement of serum level of myeloperoxidase before sternotomy and after sternal closure.

ELIGIBILITY:
Inclusion Criteria:

* ischemic heart disease

Exclusion Criteria:

* valve disease
* diabetes millitus

Ages: 30 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 336 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander S Nemkov, PhD, MD, Study Director — PSPbGMU
Locations (1):
- First Pavlov State Medical University of St. Petersburg, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 2015-2019 Location: North-West of Russia Medical clinic: Center of Cardiac Surgery of First Pavlov State Medical University
Period: Overall Study
Arm/Group | On-Pump CABG | Off-Pump CABG | BH-CABG MSC.
Started | 128 | 181 | 27
Completed | 128 | 175 | 27
Not Completed | 0 | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | On-Pump CABG | Off-Pump CABG | BH-CABG MSC. | Total
Number analyzed (Participants) | 128 | 175 | 27 | 330
Age, Continuous [Mean (Standard Deviation); unit: year] | 63.5 (7.1) | 63.5 (7.3) | 64.3 (8.95) | 64.1 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 40 | 7 | 80
  Male | 95 | 135 | 20 | 250
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 128 | 175 | 27 | 330
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 128 | 175 | 27 | 330
Ejection Fraction [Median (Inter-Quartile Range); unit: %] | 62 [59 to 66] | 62 [55 to 67] | 63 [55 to 65] | 62 [56 to 67]
troponin I [Median (Inter-Quartile Range); unit: ng/ml] | 0.014 [0.007 to 0.025] | 0.0075 [0.003 to 0.018] | 0.014 [0.0045 to 0.06] | 0.009 [0.005 to 0.02]
CRP [Median (Inter-Quartile Range); unit: g/L] — C-reactive protein
  g/L | 57.8 [55.1 to 102.3] | 5.8 [3.0 to 78.3] | 3.0 [3.0 to 7.2] | 3.0 [3 to 5.68]

OUTCOME MEASURES:

1. Primary Outcome: Myeloperoxidase
Description: Level of serum myeloperoxidase just after sternal closure
Time Frame: Level of serum myeloperoxidase just after sternal closure
Population: Patients after coronary artery bypass grafting
Measure: Median (Inter-Quartile Range); unit: g/L
Arm/Group | On-Pump CABG | Off-Pump CABG | BH-CABG MSC.
Number analyzed (Participants) | 128 | 175 | 27
g/L | 184.3 [135.01 to 250.0] | 66.5 [41.33 to 135.82] | 144.71 [95.04 to 284.92]

2. Secondary Outcome: Low Cardiac Output Syndrome
Description: Low cardiac output syndrome up to 30 days after procedure. Cardiac index (CI) was measured by invasive methods. Low cardiac output syndrome was registered when CI <2.2.
Time Frame: Up to 30 days after surgical procedure
Population: Patients with cardiac index <2.2
Measure: Count of Participants; unit: Participants
Arm/Group | On-Pump CABG | Off-Pump CABG | BH-CABG MSC.
Number analyzed (Participants) | 128 | 175 | 27
Participants | 15 | 15 | 1

3. Secondary Outcome: Length of Stay in Intensive Care Unit
Description: Length of stay in intensive care unit after operation.
Time Frame: During 30 days after procedure or more
Population: Patients after coronary artery bypass grafting
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | On-Pump CABG | Off-Pump CABG | BH-CABG MSC.
Number analyzed (Participants) | 128 | 175 | 27
days | 2 [2 to 3] | 2 [1 to 2] | 2 [2 to 5]

4. Secondary Outcome: Length of Stay in Hospital
Description: Length of stay in hospital
Time Frame: During 30 days after procedure or more
Population: Patients after coronary artery bypass grafting
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | On-Pump CABG | Off-Pump CABG | BH-CABG MSC.
Number analyzed (Participants) | 128 | 175 | 27
days | 13 [11 to 15] | 12 [10 to 13] | 13 [10 to 15]

5. Secondary Outcome: Cumulative Dose of Inotrope
Description: Calculated according: Cumulative dose of inotrope = Days dose of inotrope * days of administration of inotrope
Time Frame: Up to 30 days after procedure
Population: Patients after coronary artery bypass grafting
Measure: Median (Inter-Quartile Range); unit: mg*days
Arm/Group | On-Pump CABG | Off-Pump CABG | BH-CABG MSC.
Number analyzed (Participants) | 128 | 175 | 27
mg*days | 0 [0 to 0.12] | 0 [0 to 0.05] | 0 [0 to 1.14]

6. Secondary Outcome: Days of Administration of Inotrope
Description: Period of inotrope administration
Time Frame: During 30 days after procedure or more
Population: Patients after procedure
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | On-Pump CABG | Off-Pump CABG | BH-CABG MSC.
Number analyzed (Participants) | 128 | 175 | 27
days | 0 [0 to 2] | 0 [0 to 1] | 0 [0 to 1.5]

7. Secondary Outcome: Pulmonary Ventilation
Description: Length of pulmonary ventilation
Time Frame: During 30 days after procedure or more
Population: Patients after coronary artery bypas grafting
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | On-Pump CABG | Off-Pump CABG | BH-CABG MSC.
Number analyzed (Participants) | 128 | 175 | 27
days | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 2]

8. Secondary Outcome: Systolic Function
Description: Measured with echocardiography (Ejection Fraction)
Time Frame: Up to 14 days after surgical procedure
Population: Patients after coronary artery bypass grafting
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | On-Pump CABG | Off-Pump CABG | BH-CABG MSC.
Number analyzed (Participants) | 128 | 175 | 27
units on a scale | 62 [59 to 66] | 62 [55 to 67] | 63 [55 to 65]

9. Secondary Outcome: Diastolic Function
Description: Measured with echocardiography (End-Diastolic Volume)
Time Frame: Up to 14 days after surgical procedure
Population: Patients after CABG
Measure: Median (95% Confidence Interval); unit: ml
Arm/Group | On-Pump CABG | Off-Pump CABG | BH-CABG MSC.
Number analyzed (Participants) | 128 | 175 | 27
ml | 106.0 [81.0 to 131.0] | 97.0 [79.0 to 122.0] | 109.5 [96.0 to 136.5]

10. Secondary Outcome: Number of Participants With Reoperation
Description: Number of participants with reoperation due to cardiac complication. Cardiac complication: graft dysfunction with cardiac index<2.2.
Time Frame: Up to 30 days after procedure
Population: Patients after procedure
Measure: Count of Participants; unit: Participants
Groups:
- On-pump CABG: On-pump coronary artery bypass grafting.
- Off-pump CABG: Off-pump coronary artery bypass grafting
- Pump-assisted CABG: coronary artery bypass grafting with heart-lung machine without cross-clamping of the aorta
Arm/Group | On-pump CABG | Off-pump CABG | Pump-assisted CABG
Number analyzed (Participants) | 128 | 175 | 27
Participants | 1 | 1 | 0

11. Secondary Outcome: Renal Dysfunction
Description: Serum creatinine level after surgical operation larger than 25% level before operation
Time Frame: Perioperative (before sternotomy and after sternal closure)
Population: Patients after procedure
Measure: Count of Participants; unit: Participants
Groups:
- On-pump CABG: On-pump CABG
- Off-pump CABG: Off-pump CABG
- Pump-assisted CABG: Pump-assisted CABG
Arm/Group | On-pump CABG | Off-pump CABG | Pump-assisted CABG
Number analyzed (Participants) | 128 | 175 | 27
Participants | 70 | 49 | 7

12. Secondary Outcome: Atrial Fibrillation.
Description: New onset atrial fibrillation after operation.
Time Frame: Up to 30 days after procedure
Population: Patients after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | On-pump CABG | Off-pump CABG | Pump-assisted CABG
Number analyzed (Participants) | 128 | 175 | 27
Participants | 27 | 26 | 8

13. Other Pre Specified Outcome: Death
Description: Death after surgical procedure
Time Frame: During 30 days after procedure
Population: Patients after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | On-pump CABG | Off-pump CABG | Pump-assisted CABG
Number analyzed (Participants) | 128 | 175 | 27
Participants | 7 | 4 | 0

14. Other Pre Specified Outcome: Stroke
Description: Stroke after surgical procedure
Time Frame: During 30 days after procedure
Population: Patients after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | On-pump CABG | Off-pump CABG | Pump-assisted CABG
Number analyzed (Participants) | 128 | 175 | 27
Participants | 3 | 6 | 3

ADVERSE EVENTS:
Time Frame: 30 days follow up
Description: All-Cause Mortality: The occurrence of death due to any cause. Serious Adverse Events. 15 participants died in both the "On-pump CABG" and "Off-pump CABG" Arms/Groups.
Arm/Group | On-pump CABG | Off-pump CABG | Pump-assisted CABG
All-Cause Mortality (participants affected / at risk) | 15/128 | 15/175 | 0/27
Serious Adverse Events (participants affected / at risk) | 15/128 | 15/175 | 1/27
Other Adverse Events (participants affected / at risk) | 1/128 | 0/175 | 1/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | On-pump CABG (N=128) | Off-pump CABG (N=175) | Pump-assisted CABG (N=27)
Low cardiac output synfrome (Cardiac disorders) | 15 (15) | 15 (15) | 1 (1) — Low cardiac output synfrome when cardiac index <2.2
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | On-pump CABG (N=128) | Off-pump CABG (N=175) | Pump-assisted CABG (N=27)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Unequal amount of participants in arms (few patients were enrolled in off-pump arm).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT03050489/Prot_SAP_000.pdf